CLINICAL TRIAL: NCT00375427
Title: A Prospective, Randomized, Multi-center Comparative 2-arm Trial of Efficacy and Safety of Zoledronic Acid (Every 3-months vs. Every 4 Weeks) Beyond Approximately 1 Year of Treatment With Zoledronic Acid in Patients With Bone Lesions From Breast Cancer
Brief Title: Safety and Efficacy of Zoledronic Acid in Patients With Breast Cancer With Metastatic Bone Lesions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446EIT14
Record Dates: First submitted 2006-09-12; First posted 2006-09-13 (Estimated); Results first posted 2011-08-04 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2011-07

CONDITIONS: Breast Cancer With Bone Metastasis
Keywords: Breast cancer; Zoledronic acid; Skeletal related events (SRE)
MeSH Terms: conditions — Breast Neoplasms | interventions — Zoledronic Acid

ARMS (2):
- Every 3 months (Experimental): Zoledronic acid as a 15-minute (at least) intravenous (i.v.) infusion every three months. The dose of study drug will be the same administered before the study entry, that is 4 mg or a reduced dose, i.e. 3.5 mg, or 3.3 mg or 3.0 mg. Randomized patients will receive a maximum of 4 infusions in this group.
  Interventions: Drug: Zoledronic acid
- Every 4 weeks (Experimental): Zoledronic acid as a 15-minute (at least) intravenous (i.v.) infusion every 4 weeks. The dose of study drug will be the same administered before the study entry, that is 4 mg or a reduced dose, i.e. 3.5 mg, or 3.3 mg or 3.0 mg. Patients randomized to this group will receive up to 12 infusions.
  Interventions: Drug: Zoledronic acid

INTERVENTIONS:
Drug: Zoledronic acid — Zoledronic acid as a 15-minute (at least) intravenous (i.v.) infusion. The dose of study drug will be the same administered before the study entry, that is 4 mg or a reduced dose, i.e. 3.5 mg, or 3.3 mg or 3.0 mg.
  Other Names: ZOL446; Zometa®

SUMMARY:
The objective of this study is to assess the clinical benefit of two different dosing schedules of zoledronic acid in patients with metastatic bone lesions from breast cancer who have already been treated with zoledronic acid for about one year.

ELIGIBILITY:
Inclusion criteria:

* Female patients ≥ 18 years of age.
* Written informed consent given.
* Histologically confirmed Stage IV breast cancer with at least one bone metastasis radiologically confirmed.
* Previous treatment with zoledronic acid every 3-4 weeks, for 9-12 infusions over no more than 15 months.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2 .
* Life expectancy ≥ 1 year.

Exclusion criteria:

* More than 3 months since last infusion of Zoledronic Acid (Zometa®).
* Treatments with other bisphosphonate than Zoledronic Acid (Zometa®) at any time prior to study entry.
* Serum creatinine > 3 mg/dL (265 μmol/L) or calculated (Cockcroft-Gault formula) creatinine clearance (CLCr) < 30 mL/min CrCl = ({[140-age (years)] x weight(kg)}/ [72 x serum creatinine (mg/dL)])x 0.85
* Corrected (adjusted for serum albumin) serum calcium < 8 mg/dl (2 mmol/L) or > 12 mg/dL ( 3.0 mmol/L).
* Current active dental problem including infection of the teeth or jawbone (maxilla or mandibular); dental or fixture trauma, or a recurrent or prior diagnosis of osteonecrosis of the jaw (ONJ), of exposed bone in the mouth, or of slow healing after dental procedures.
* Recent (within 6 weeks) or planned dental or jaw surgery (e.g. extraction, implants).
* Pregnant patients (with a positive pregnancy test prior to study entry) or lactating patients. Women of childbearing potential not using effective methods of birth control (e.g. abstinence, oral contraceptives or implants, IUD, vaginal diaphragm or sponge, or condom with spermicide).
* History of non-compliance to medical regimens or potential unreliable behavior.
* Known sensitivity to study drug(s) or class of study drug(s).
* Patients with severe medical condition(s) that in the view of the investigator prohibits participation in the study
* Use of any other investigational agent in the last 30 days.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2006-02; Primary Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Forlì, Italy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total enrollment was 430; five participants were screened but not treated.
Groups:
- Zoledronic Acid Every 3 Months: Zoledronic acid given as a 15-minute (at least) i.v. infusion every three months. The dose of study drug was the same as administered before study entry; that is, 4 mg or a reduced dose, i.e. 3.5 mg, or 3.3 mg or 3.0 mg. Randomized participants received a maximum of 4 infusions in this group.
- Zoledronic Acid Every 4 Weeks: Zoledronic acid given as a 15-minute (at least) i.v. infusion every 4 weeks. The dose of study drug was the as same administered before study entry; that is, 4 mg or a reduced dose, i.e. 3.5 mg, or 3.3 mg or 3.0 mg. Participants randomized to this group received up to 12 infusions.
Period: Overall Study
Arm/Group | Zoledronic Acid Every 3 Months | Zoledronic Acid Every 4 Weeks
Started | 209 (Total enrollment was 430 but five patients were screened but not treated.) | 216
Completed | 149 | 142
Not Completed | 60 | 74
Not completed — Adverse Event | 21 | 27
Not completed — Abnormal test procedure result(s) | 0 | 1
Not completed — Abnormal laboratory value(s) | 1 | 2
Not completed — Unsatisfactory therapeutic effect | 4 | 4
Not completed — Patient no longer requires study drug | 3 | 7
Not completed — Protocol Violation | 10 | 8
Not completed — Withdrawal by Subject | 9 | 13
Not completed — Lost to Follow-up | 1 | 1
Not completed — Administrative reasons | 0 | 1
Not completed — Death | 11 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zoledronic Acid Every 3 Months | Zoledronic Acid Every 4 Weeks | Total
Number analyzed (Participants) | 209 | 216 | 425
Age Continuous [Mean (Standard Deviation); unit: years] | 60.4 (11.9) | 59.8 (11.8) | 60.1 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 209 | 216 | 425
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Annual Overall Skeletal Morbidity Rate (SMR)
Description: The SMR was computed by summing all Skeletal Related Event(s) (SREs)which occurred during the observation period and dividing it by the ratio "days of observation period / 365.25", for each participant. SRE was defined as: pathologic bone fracture, spinal cord compression, surgery to bone both curative and prophylactic, radiation therapy to bone, or hypercalcemia of malignancy.
  SMR (years) = 365.25 x SMR(days) where SMR (days) = total number of SREs / total SRE risk period (days). Risk period for SMR was computed as the days from randomization date to the date of last visit.
Time Frame: 12 months
Population: Intent-to-treat (ITT) population will include all randomized patients.
Measure: Mean (Standard Deviation); unit: Number of Skeletal Events per Year
Arm/Group | Zoledronic Acid Every 3 Months | Zoledronic Acid Every 4 Weeks
Number analyzed (Participants) | 209 | 216
Number of Skeletal Events per Year | 0.26 (0.81) | 0.22 (0.57)

2. Secondary Outcome: Percentage of Participants Experiencing Skeletal Related Event(s) (SREs)
Description: Skeletal Related Events (SREs) are defined as a:
  * pathologic bone fracture such as non-vertebral and vertebral compression fractures
  * spinal cord compression identified by positive diagnosis documented by X-ray evidence
  * surgery to bone both curative and prophylactic
  * radiation therapy to bone including palliative, therapeutic or prophylactic
  * hypercalcemia of malignancy, defined as a corrected serum calcium > 12 mg/dl (3.00 mmol/l) or a lower level of hypercalcemia which is symptomatic and which requires active treatment other than rehydration.
Time Frame: 12 month
Population: Intent-to-treat (ITT) population will include all randomized patients.
Measure: Number; unit: Percentage of Participants
Arm/Group | Zoledronic Acid Every 3 Months | Zoledronic Acid Every 4 Weeks
Number analyzed (Participants) | 209 | 216
Percentage of Participants
  Patient with any SRE | 14.83 | 15.28
  Vertebral pathological fracture | 1.44 | 1.85
  Non vertebral pathological fracture | 3.35 | 2.31
  Spinal cord compression | 0.96 | 0.46
  Radiation to bone | 10.53 | 11.11
  Surgery to bone | 0.96 | 0.46
  Hypercalcemia of malignancy | 0.48 | 1.85

3. Secondary Outcome: Annual Incidence of Any Skeletal Related Events (SREs)
Description: Skeletal Related Events (SREs) are defined as a:
  * pathologic bone fracture such as non-vertebral and vertebral
  * spinal cord compression identified by X-rays evidence
  * surgery to bone both curative and prophylactic
  * radiation therapy to bone including palliative, therapeutic or prophylactic
  * hypercalcemia of malignancy, defined as a corrected serum calcium > 12 mg/dl (3.00 mmol/l) or a lower level of hypercalcemia which is symptomatic and which requires active treatment other than rehydration. Annual incidence for each SRE was computed in the same way as annual overall SMR.
Time Frame: 12 months
Population: Intent-to-treat (ITT) population will include all randomized patients.
Measure: Mean (Standard Deviation); unit: Number of SRE per Year
Arm/Group | Zoledronic Acid Every 3 Months | Zoledronic Acid Every 4 Weeks
Number analyzed (Participants) | 209 | 216
Number of SRE per Year
  Vertebral pathological fracture rate | 0.02 (0.19) | 0.02 (0.15)
  Non-vertebral pathological fracture rate | 0.08 (0.58) | 0.03 (0.20)
  Spinal cord compression rate | 0.01 (0.10) | 0.00 (0.07)
  Radiation to bone rate | 0.17 (0.67) | 0.14 (0.43)
  Surgery to bone rate | 0.02 (0.21) | 0.00 (0.07)
  Hypercalcemia of malignancy rate | 0.01 (0.08) | 0.02 (0.16)

4. Secondary Outcome: Median Time to First Skeletal Related Event(s) (SRE)
Description: Median Time to first skeletal related event (SRE) is defined as the time from randomization to the date of first occurrence of any SRE which includes at least one of the following: radiation therapy to bone, pathologic bone fracture, spinal cord compression, surgery to bone, and hypercalcemia of malignancy (HCM). Due to the few numbers of SRE, Kaplan-Meier estimate never reaches a failure probability >=25%; so median time, 25th and 75th percentiles are not determined.For this reason only the estimated percentage of patient SRE free are reported at each time point.
Time Frame: 12 month
Measure: Number; unit: Day
Arm/Group | Zoledronic Acid Every 3 Months | Zoledronic Acid Every 4 Weeks
Number analyzed (Participants) | 209 | 216
Day | NA — NA=Not evaluable. Due to the low incidence of SRE, K-M estimates never reach a failure probability ≥25%; so median time, 25th and 75th percentiles aren't determined. Time can't be estimated because of insufficient SRE to reach the quartiles | NA — NA=Not evaluable. Due to the low incidence of SRE, K-M estimates never reach a failure probability ≥25%; so median time, 25th and 75th percentiles aren't determined. Time can't be estimated because of insufficient SRE to reach the quartiles

5. Secondary Outcome: Percentage of Participants Skeletal Related Event (SRE) Free
Description: Percentage of participants SRE free is defined as the Kaplan-Meier estimate of participants free of any Skeletal Related Events(SRE) at each time point.
  Skeletal Related Events (SREs) are:
  * pathologic bone fracture; non-vertebral and vertebral
  * spinal cord compression identified by X-rays
  * surgery to bone both curative and prophylactic
  * radiation therapy to bone (palliative, therapeutic or prophylactic)
  * hypercalcemia of malignancy, defined as a corrected serum calcium > 12 mg/dl (3.00 mmol/l) or a lower level which is symptomatic and requires treatment other than rehydration.
Time Frame: 12 months
Population: Intent-to-treat (ITT) population will include all randomized patients.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zoledronic Acid Every 3 Months | Zoledronic Acid Every 4 Weeks
Number analyzed (Participants) | 209 | 216
Percentage of participants
  At Month 1 | 99 [96 to 100] | 98 [95 to 99]
  At Month 2 | 98 [94 to 99] | 98 [94 to 99]
  At Month 3 | 96 [92 to 98] | 97 [93 to 98]
  At Month 4 | 94 [90 to 97] | 95 [91 to 97]
  At Month 5 | 94 [89 to 96] | 93 [89 to 96]
  At Month 6 | 93 [89 to 96] | 92 [87 to 95]
  At Month 7 | 88 [83 to 92] | 90 [85 to 93]
  At Month 8 | 86 [80 to 90] | 88 [83 to 92]
  At Month 9 | 85 [79 to 90] | 85 [79 to 89]
  At Month 10 | 84 [78 to 89] | 83 [77 to 88]
  At Month 11 | 83 [77 to 88] | 83 [77 to 88]
  At Month 12 | 78 [63 to 87] | 82 [75 to 87]

6. Secondary Outcome: Composite Bone Pain Score According to the Brief Pain Inventory (BPI) Questionnaire
Description: Bone pain was assessed by means of a pain score obtained using the Brief Pain Inventory (BPI) questionnaire. The BPI can produce three pain scores: worst pain, a composite pain score, and a pain interference score. The composite pain score, which is the average of questions 3, 4, 5 and 6 of the questionnaire was used in this study. Pain was rated on a scale of 0 (no pain) to 10 (pain as bad as you can imagine). The outcome is given as the median score for participants at baseline, and 3, 6, 9 and 12 months of treatment
Time Frame: At Baseline, Month 3, Month 6, Month 9 and Month 12
Population: Intent-to-treat (ITT) population will include all randomized patients. All ITT patients with BPI questionnaire filled up at baseline were included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Zoledronic Acid Every 3 Months | Zoledronic Acid Every 4 Weeks
Number analyzed (Participants) | 186 | 185
score on a scale
  Baseline (N= 186, 185) | 2.0 (1.8) | 2.1 (1.9)
  Month 3 (N= 156, 163) | 2.3 (2.0) | 2.2 (1.9)
  Month 6 (N= 143, 160) | 2.3 (2.2) | 1.9 (1.8)
  Month 9 (N= 131, 130) | 2.3 (2.2) | 2.1 (2.0)
  Month 12 (N= 135, 124) | 2.4 (2.3) | 2.1 (2.0)

7. Secondary Outcome: Evaluation of Pain According to Verbal Rating Scale (VRS) Based on Median Score Value
Description: Pain intensity at rest and on movement is rated by the patient by means of a validated 6-point Verbal Rating Scale (VRS) and refers to the pain which occurred during the last week before the assessment. Median score value is the median of all the observed scores (none=0, very mild=1, mild=2, moderate=3, severe=5 and very severe=6) at each time point.
Time Frame: At Baseline, Month 3, Month 6, Month 9 and Month 12
Population: Intent-to-treat (ITT) population will include all randomized patients.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Zoledronic Acid Every 3 Months | Zoledronic Acid Every 4 Weeks
Number analyzed (Participants) | 209 | 216
score on a scale
  At Rest: Baseline | 1 [1.00 to 5.00] | 1 [1.00 to 6.00]
  At Rest: Month 3 | 2 [1.00 to 6.00] | 2 [1.00 to 5.00]
  At Rest: Month 6 | 2 [1.00 to 5.00] | 1 [1.00 to 6.00]
  At Rest: Month 9 | 1 [1.00 to 5.00] | 1 [1.00 to 5.00]
  At Rest: Month 12 | 2 [1.00 to 6.00] | 1 [1.00 to 6.00]
  At Movement : Baseline | 2 [1.00 to 5.00] | 2 [1.00 to 6.00]
  At Movement : Month 3 | 2 [1.00 to 6.00] | 2 [1.00 to 6.00]
  At Movement : Month 6 | 2 [1.00 to 6.00] | 2 [1.00 to 6.00]
  At Movement : Month 9 | 2 [1.00 to 6.00] | 2 [1.00 to 6.00]
  At Movement : Month 12 | 2.5 [1.00 to 6.00] | 2 [1.00 to 6.00]

8. Secondary Outcome: Use Of Analgesic Medications According to the Analgesic Score Scale
Description: The analgesic score used for this study is modified from the Radiation Therapy Oncology Group (RTOG) analgesic score scale. The scale represents type of medication administered from 0 to 4 where:
  0 = None
  1. = Minor analgesics (aspirin, NSAID, acetaminophen, propoxyphene, etc.)
  2. = Tranquilisers, antidepressants, muscle relaxants, and steroids
  3. = Mild narcotics (oxycodone, meperidine, codeine, etc.)
  4. = Strong narcotics (morphine, hydromorphone, etc.) The outcome is given a the median score for the participants at Baseline and 3, 6, 9 and 12 months of treatment
Time Frame: At Baseline, Month 3, Month 6, Month 9 and Month 12
Population: Intent-to-treat (ITT) population will include all randomized patients.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Zoledronic Acid Every 3 Months | Zoledronic Acid Every 4 Weeks
Number analyzed (Participants) | 209 | 216
score on a scale
  Baseline | 0 [0 to 4] | 0 [0 to 4]
  Month 3 | 0 [0 to 4] | 0 [0 to 4]
  Month 6 | 0 [0 to 4] | 0 [0 to 4]
  Month 9 | 0 [0 to 4] | 0 [0 to 4]
  Month 12 | 0 [0 to 4] | 0 [0 to 4]

9. Secondary Outcome: Assessment of the Eastern Cooperative Oncology Group (ECOG) Performance Score
Description: ECOG Performance Score has 4 grades. 0 = Fully active, able to carry out all pre-disease activities; 1 = Restricted in strenuous activity but ambulatory and able to carry out work of light or sedentary nature; 2 = Ambulatory and capable of all self-care but unable to carry out work activities. Active about 50% of waking hours; 3 = Capable of limited self-care, confined to bed/chair more than 50% of waking hours; 4 = Completely disabled; cannot carry on self-care. Totally confined to bed/chair. Outcome is given as median score for participants at Baseline and 3, 6 , 9 and 12 months of treatment
Time Frame: At Baseline, Month 3, Month 6, Month 9 and Month 12
Population: Intent-to-treat (ITT) population will include all randomized patients.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Zoledronic Acid Every 3 Months | Zoledronic Acid Every 4 Weeks
Number analyzed (Participants) | 209 | 216
score on a scale
  Baseline | 0 [0 to 2] | 0 [0 to 2]
  Month 3 | 0 [0 to 3] | 0 [0 to 3]
  Month 6 | 0 [0 to 2] | 0 [0 to 2]
  Month 9 | 0 [0 to 2] | 0 [0 to 2]
  Month 12 | 0 [0 to 4] | 0 [0 to 4]

ADVERSE EVENTS:
Arm/Group | Zoledronic Acid Every 3 Months | Zoledronic Acid Every 4 Weeks
Serious Adverse Events (participants affected / at risk) | 21/209 | 29/216
Other Adverse Events (participants affected / at risk) | 133/209 | 161/216
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid Every 3 Months (N=209) | Zoledronic Acid Every 4 Weeks (N=216)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 2
Mucosal inflammation (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1
Acute sinusitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 2 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Jaw disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 4 | 3
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cranial nerve paralysis (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 1
Paraparesis (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Sopor (Psychiatric disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Breast operation (Surgical and medical procedures) | 1 | 0
Laparoscopic surgery (Surgical and medical procedures) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid Every 3 Months (N=209) | Zoledronic Acid Every 4 Weeks (N=216)
Anaemia (Blood and lymphatic system disorders) | 13 | 21
Neutropenia (Blood and lymphatic system disorders) | 11 | 18
Vertigo (Ear and labyrinth disorders) | 2 | 11
Abdominal pain (Gastrointestinal disorders) | 12 | 15
Abdominal pain upper (Gastrointestinal disorders) | 16 | 20
Constipation (Gastrointestinal disorders) | 12 | 15
Diarrhoea (Gastrointestinal disorders) | 12 | 17
Nausea (Gastrointestinal disorders) | 24 | 32
Vomiting (Gastrointestinal disorders) | 13 | 21
Asthenia (General disorders) | 18 | 33
Fatigue (General disorders) | 10 | 12
Pain (General disorders) | 10 | 15
Pyrexia (General disorders) | 22 | 28
Gamma-glutamyltransferase increased (Investigations) | 8 | 12
Anorexia (Metabolism and nutrition disorders) | 5 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 13
Bone pain (Musculoskeletal and connective tissue disorders) | 56 | 64
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 12
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 67 | 68
Headache (Nervous system disorders) | 14 | 15
Paraesthesia (Nervous system disorders) | 11 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 13
Rash (Skin and subcutaneous tissue disorders) | 3 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.